CLINICAL TRIAL: NCT07095439
Title: Efficacy and Toxicity of Total Neoadjuvant Sandwich Treatment Via Short Course Radiotherapy in the Treatment of Stage II and III Rectal Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD200/2023
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Short course radiotherapy; Total neoadjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total neoadjuvant treatment via short course radiotherapy (Experimental): Participants in this arm receive 4 cycles of induction chemotherapy CAPEOX (or 5 cycles of FOLFOX6), followed by short course radiotherapy (25 Gy in 5 fractions) delivered via IMRT technique ,then consolidation chemotherapy in the form of : 2 cycles of CAPOX (or, 4 cycles of FOLFOX6). Total mesorectal excision (TME) will be performed for non-metastatic patients within 8-12 weeks of the short course radiotherapy.
  Interventions: Radiation: Total Neoadjuvant Treatment

INTERVENTIONS:
Radiation: Total Neoadjuvant Treatment — Participants in this arm receive 4 cycles of induction chemotherapy CAPEOX (or 5 cycles of FOLFOX6), followed by short course radiotherapy (25 Gy in 5 fractions) delivered via IMRT technique ,then consolidation chemotherapy in the form of : 2 cycles of CAPOX (or, 4 cycles of FOLFOX6). Total mesorectal excision (TME) will be performed for non-metastatic patients within 8-12 weeks of the short course radiotherapy.
  Other Names: Short course radiotherapy

SUMMARY:
Several trials showed that total neoadjuvant treatment (TNT) in stage II/III rectal cancer patients had better outcomes when compared with standard neoadjuvant long-course radiotherapy (CRT). Recently, based on the RAPIDO and POLISH II trials a short course radiotherapy (SCRT)-including TNT strategy had better oncologic outcomes and comparable toxicities. Moreover, cost-effectively, an SCRT-including TNT strategy is more convenient than a CRT-based TNT approach. In addition, systemic chemotherapy is often used to treat occult or micrometastatic disease in intermediate and locally advanced rectal cancer. However, the timing of chemotherapy delivery remains a topic of debate. In this context, and since rapid access to radiotherapy treatment is limited, especially in developing countries, a TNT strategy whereby adjuvant chemotherapy is replaced by systemic chemotherapy delivered before and after SCRT according to a "sandwich" treatment can avoid delays in treatment start with equivalent outcomes.

DETAILED DESCRIPTION:
Rectal cancer is a common malignancy that often requires multimodal treatment approaches for optimal outcomes. Neoadjuvant chemoradiotherapy is a standard of care for stage II-III rectal cancer, with total neoadjuvant treatment (TNT) being an emerging strategy. Long-course chemoradiotherapy (CRT) and short-course radiotherapy (SCRT) are both commonly used as neoadjuvant treatments for stage II-III rectal cancer. SCRT consists of 5 fractions of 5 Gy followed by surgery, which can be performed 1 to 8 weeks later [1-3]. Studies have shown that both approaches have similar survival rates, toxicity levels, and patient-reported outcomes [4-6].

The Uppsala trial was the starting point for the acceptance of preoperative SCRT [7], with the Stockholm I trial running in parallel [8]. The subsequent Swedish Rectal Cancer Trial, which randomized patients between surgery alone and preoperative SCRT, showed not only improved local control but also a survival benefit [9]. Although criticism was raised regarding the quality of surgery performed in these trials, the Dutch TME trial confirmed that preoperative SCRT improved local control, with certain subgroups showing a survival benefit [10,11]. Randomized data also suggest that SCRT should be preferred in resectable rectal cancer, as it leads to decreased short-term toxicity and no differences in long-term oncologic outcomes and late toxicity compared to preoperative CRT [12].

The risk of developing metachronous metastases in intermediate and locally advanced rectal cancer is high (25-65%), and systemic chemotherapy aims to treat the occult or micrometastatic disease that may later appear as distant metastases [13-15]. However, there are at least two arguments against postoperative delivery of chemotherapy. Firstly, rectal cancer surgery is associated with a substantial risk of postoperative complications that may prevent patients from tolerating postoperative chemotherapy [16,17]. Secondly, in the early stages of the disease when microscopic dissemination is limited, systemic chemotherapy would theoretically be expected to be most effective. Additionally, surgery, particularly if extensive, may accelerate tumor growth [18,19].

Recent studies have shown promising results with a strategy of delivering preoperative SCRT followed by delayed surgery [20-22]. Moreover, (SCRT)-including TNT strategy was investigated in several large trials. A Dutch phase II trial has reported high response rates and radical resection in patients with resectable metastatic rectal cancer who received SCRT followed by preoperative chemotherapy including bevacizumab [23]. The Polish II study included patients with locally advanced rectal cancer and compared preoperative SCRT followed by chemotherapy with CRT. They reported decreased acute toxicities and better overall survival (OS) [24]. Additionally the RAPIDO trial has concluded that SCRT followed by preoperative chemotherapy showed lower risk of disease related treatment failure and comparable toxicity profile when compared with preoperative CRT [25].

The above mentioned factors highlight the need for effective neoadjuvant treatment strategies that incorporate systemic chemotherapy and minimize the risk of postoperative complications. Two trials have explored the use of TNT using CRT where chemotherapy is delivered before and after radiotherapy (via a sandwich technique), one trial offered adjuvant chemotherapy as well. Both trials showed that neoadjuvant CRT based sandwich technique is well tolerated and highly effective in terms of PCR rate [26-27].

The timing of chemotherapy delivery remains a topic of debate, with concerns over postoperative complications. Both SCRT and CRT have been shown to have similar efficacy and safety profiles, SCRT has gained acceptance as a preferred option due to its decreased short-term toxicity and similar long-term outcomes. Moreover access to radiotherapy treatment in some developing countries can be limited, leading to delays in treatment initiation [28]. In this setting a TNT strategy utilizing systemic chemotherapy delivered before and after SCRT (known as a "sandwich" treatment) could provide equivalent outcomes while avoiding delays in treatment initiation and being more cost-effective compared to a CRT-based TNT approach.

The primary end point is to assess the rate of pathological complete response (pCR) after total mesorectal excision (TME). The secondary end points are to explore radiotherapy-related toxicities, post-operative complications and median disease free survival of systemic chemotherapy delivered before and after short course radiotherapy (SCRT) according to a "sandwich" technique.

ELIGIBILITY:
Inclusion Criteria:

* · Patients aged 18 years old till 70 years old.

  * Pathologically confirmed rectal adenocarcinoma of low or mid rectum (less than 16 cm from the anal verge on endoscopy)
  * Stage II and stage III by imaging (T3 N any M0 or T1-2 N+ve M0) [29]; staged with MRI rectal protocol or EUS.
  * The disease was staged with CT imaging of chest, abdomen and pelvis pretreatment.
  * Eastern Cooperative Oncology Group (ECOG) performance status= 0-2.
  * The following laboratory results are required: absolute neutrophilic count of 1.5 × 10⁹ cells per L or higher, platelet count of 100 × 10⁹ per L or higher, a clinically acceptable haemoglobin level, a creatinine level indicating renal clearance of 50 mL/min or higher, and bilirubin level below 2 mg/dL.
  * Written informed consent.

Exclusion Criteria:

* · Previous surgical treatment for rectal cancer or concurrent fistulising inflammatory bowel disease of the rectum.

  * Surgical or medical inoperability.
  * Previous pelvic radiotherapy.
  * Second malignancy within the last 5 years.
  * Patients with diseases that do not allow receipt of chemotherapy or radiotherapy as grade 3 neuropathy and severe cardiovascular disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 6 months, from induction chemotherapy till total mesorectal excision
  The complete disappearance of all signs of cancer in tissue samples after treatment with chemotherapy and radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled M Abdel Karim, MD, Principal Investigator — Faculty of medicine, Ain Shams University; Nesreen A Mosalam, MD, Study Director — Faculty of medicine, Ain Shams University; Lamiaa M Ahmed, MD, Study Director — Faculty of medicine, Ain Shams University; Sara E Zaki, MD, Study Director — Faculty of medicine, Ain Shams University
Locations (1):
- Clinical oncology and nuclear medicine Department, Faculty of medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Because the study is conducted within an academic setting and involves patient data that cannot be shared publicly due to confidentiality and ethical considerations